CLINICAL TRIAL: NCT06605105
Title: A Phase III Long-Term Extension Trial With Optional Additional Doses of CYB003 to Assess the Safety and Long-term Efficacy in Participants With Major Depressive Disorder (EXTEND)
Brief Title: Phase III Long-term Extension Trial to Assess Safety and Efficacy of CYB003 in MDD (EXTEND)
Acronym: EXTEND
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cybin IRL Limited (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYB003-004
Record Dates: First submitted 2024-09-16; First posted 2024-09-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Psilocybin; Psychedelic; CYB003; Depression; CYB003-002; Long-Term Extension; CYB003-003
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CYB003 (Experimental): Initial non-responders in CYB003-002 APPROACH and CYB003-003 EMBRACE, or initial responders who later relapse will be eligible to receive 16 mg of CYB003 in 2 of 2 medicine sessions, approximately three weeks apart. If a participant relapses again, the participant may receive an additional single 16mg of CYB003 (maximum of 3 16mg doses in CYB003-004 EXTEND). Participants will continue on their current antidepressants and receive psychological support throughout the study.
  Interventions: Drug: CYB003

INTERVENTIONS:
Drug: CYB003 — CYB003 is a deuterated psilocin analog

SUMMARY:
This is a long- term extension of the double-blind trials APPROACH (CYB003-002) and EMBRACE (CYB003-003). Its aim is to examine the safety and long-term efficacy of CYB003 in participants with MDD.

ELIGIBILITY:
Inclusion Criteria:

* Has successfully completed either CYB003-002 APPROACH or CYB003-003 EMBRACE and received both dose administrations of trial medication
* Has continued the same antidepressant medication at the stable dose/day throughout CYB003-002 APPROACH or CYB003-003 EMBRACE
* Has provided written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form
* Participants capable of producing sperm must use a condom plus spermicide (where publicly available) during the trial and for 12 weeks after their final dose of IP, if their partner is a person of childbearing potential. In addition, their partner of childbearing potential must continue to use a highly effective method of contraception (i.e., failure rate less than 1% when used consistently and correctly) throughout the trial until 12 weeks after the participant's final dose of IP
* Participants of childbearing potential (POCBP) who have a partner capable of producing sperm must agree to continue to use a highly effective method of contraception (i.e., failure rate of less than 1% when used consistently and correctly) in combination with the use of a condom plus spermicide (where publicly available) during the trial and for 12 weeks after their final dose of IP
* Female participants must have a negative pregnancy test at Baseline (the end of trial [EOT] Visit in the APPROACH or EMBRACE trial), and prior to dose administration on the dosing day

Exclusion Criteria:

* newly developed symptoms of schizophrenia spectrum or other psychotic disorders that manifested in the APPROACH or EMBRACE trial
* Significant suicide risk as defined by suicidal ideation as endorsed on items 4 or 5 on the C-SSRS at Baseline OR has experienced an adverse event (AE) of suicide ideation/attempt or self-harm in CYB003-002 APPROACH OR has had a >1 point change in item 1 or 2 of the C-SSRS from Screening in CYB003-002 APPROACH
* Clinically relevant arrhythmia or vital sign changes noted during any of the dosing sessions in the APPROACH or EMBRACE trial
* Presence of clinically significant ECG abnormalities noted during the APPROACH or EMBRACE trials or at the Baseline of EXTEND
* Sensitivity or suspected sensitivity to CYB003 noted in the APPROACH or EMBRACE trial
* Positive urine test for drugs of abuse, or alcohol breath test prior to dosing.
* Unwilling to consent to audio and video recording of psychological support and dosing sessions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, Day 28, Day 56, Day 84, Day 112, Day 140, Day 168, Day 196, Day 244, Day 252, Day 280, Day 301; additional assessments at Day -15, Day -1, Day 2, Day 10, Day 17, Day 21, Day 23, Day 31, Day 42 if non-response or relapse criteria met
  The MADRS is a 10-item scale with ratings based on a clinical interview which moves from broadly phrased questions about symptoms to more detailed ones allowing a precise rating of severity. The scale consists of ten items rated on a scale from 0 to 6, resulting in a total score ranging from 0 (normal / symptom absent) to 60 (severe depression).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Chair — Cybin IRL Limited
Locations (10):
- United States (10):
  - Open Mind Collective / UCSF Medical Center - Mount Zion, San Francisco, California
  - Research Centers of America, Hollywood, Florida
  - Segal Trials Center for Psychedelic Research, Lauderhill, Florida
  - Cenexel iResearcvh Atlanta, LLC, Atlanta, Georgia
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Sunstone Medical, PC, Rockville, Maryland
  - Adams Clinical, Watertown, Massachusetts
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Cedar Clinical Research, Draper, Utah

IPD SHARING:
Plan to Share IPD: No